CLINICAL TRIAL: NCT04615533
Title: Validity Reliability of FrailBESTest in Older Adults
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal Investigator, Kırıkkale University
Other Study IDs: Frail'BESTest
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Frail Elderly Syndrome; Balance; Distorted; Assessment, Self
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail older adults, assessment: Frail older adults, assessment Frail'BESTest, Clinical Frailty Scale, Mini BESTest, Berg Balance Scale, Tinetti Blance and Gait Scale
  Interventions: Other: Frail older adults, assessment

INTERVENTIONS:
Other: Frail older adults, assessment — Frail'BESTest, Clinical Frailty Scale, Mini BESTest, Berg Balance Scale, Tinnetti Balance and gait sacale

SUMMARY:
Fraility; It is an age-related biological syndrome. It is characterized by decreased resistance to stressors due to changes in functional reserves and physiological systems.

BESTest, which is frequently used in the literature, was modified and Frail'BESTest was developed to detect balance problems in fragile individuals. The test consists of 6 subtitles. These are participation, reaction, movement ability, sensory organization, biomechanical constraints, gait symmetry. When looking at the literature, the Turkish version of Frail'BESTest has not been found. For this reason, the aim of study is to examine the validity and reliability of the Turkish version of Frail'BESTest in elderly individuals and to question the effectiveness of its clinical use and to bring it to the use of other researchers.

DETAILED DESCRIPTION:
Fraility; It is an age-related biological syndrome. It is characterized by decreased resistance to stressors due to changes in functional reserves and physiological systems.Especially, the increase in the incidence of falls, loss of mobility, dependence in basic life activities, increase in hospitalizations and increased incidence of death make the diagnosis and treatment of frailty important in elderly individuals.

BESTest, which is frequently used in the literature, was modified and Frail'BESTest was developed to detect balance problems in fragile individuals. The test consists of 6 subtitles. These are participation, reaction, movement ability, sensory organization, biomechanical constraints, gait symmetry. When looking at the literature, the Turkish version of Frail'BESTest has not been found. For this reason, the aim of study is to examine the validity and reliability of the Turkish version of Frail'BESTest in elderly individuals and to question the effectiveness of its clinical use and to bring it to the use of other researchers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,

  * Your willingness to participate in research Elderly individuals with a diagnosis of frailty
  * No cooperation and communication problems

Exclusion Criteria:

* Individuals with neurological and orthopedic problems Uncontrollable hypertension

  * Those with cardiac disease
  * Those with cooperation and communication problems

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals aged 65 and over, Volunteering to participate in research, No cooperation and communication problem
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Frail'BESTest | Day 1
  The test consists of 6 subtitles. These are participation, reaction, movement ability, sensory organization, biomechanical constraints, gait symmetry.
Clinical Frailty Scale | Day 1
  Scale evaluates physical weaknesses such as comorbidity, cognitive impairment, and disability. Scale scoring is from 1 (very favorable) to 9 (terminally ill)
Mini BESTest | Day 1
  The Mini-BESTest consists of 14 items and evaluates 4 different components of dynamic balance (1) antispatient postural adjustments, (2) reactive postural control, (3) sensory orientation and (4) dynamic walking).
Berg Balance Test | Day 1
  The BBS consists of 14 items to directly monitor the maintenance of body balance during performance
Tinetti Balance and Gait Test | Day 1
  In the test used to evaluate balance, walking score is maximum 12 points, balance score is maximum 16 points and a total of 28 points

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Abit Kocaman, Principal Investigator — Kırıkkale University
Locations (1):
- Ayşe Abit Kocaman, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kubicki A, Brika M, Coquisart L, Basile G, Laroche D, Mourey F. The Frail'BESTest. An Adaptation of the "Balance Evaluation System Test" for Frail Older Adults. Description, Internal Consistency and Inter-Rater Reliability. Clin Interv Aging. 2020 Jul 30;15:1249-1262. doi: 10.2147/CIA.S247332. eCollection 2020. PMID 32801673